CLINICAL TRIAL: NCT01363570
Title: Evaluation of Wet Age-Related Macular Degeneration (AMD) Genetic Profile Interactions With Ranibizumab Treatment Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian National Institute for the Blind (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMDgene12011
Record Dates: First submitted 2011-05-30; First posted 2011-06-01 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: Age Related Macular Degeneration
Keywords: Macular Degeneration; Age related macular degeneration; Macula Risk; Genetic test; Anti-inflammatory; Anti-vascular endothelial growth factor (Anti-VEGF); Lucentis; Ranibizumab; Vision loss
MeSH Terms: conditions — Macular Degeneration; Vision Disorders | interventions — Ranibizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ranibizumab (Other): Ranibizumab is the current gold standard treatment for wet age-related macular degeneration. This intervention is approved by Health Canada, covered by OHIP (Ontario Health Insurance Plan) and used regularly by ophthalmologists in Canada. Participants will receive intravitreal injections of ranibizumab each month for up to 6 months, with ocular testing at each appointment as prescribed by the study protocol.
  Interventions: Drug: Ranibizumab

INTERVENTIONS:
Drug: Ranibizumab — Intra-vitreal injections of 0.5mg/0.05 mL dosage, injected at months 0, 1, and 2. For those requiring additional injections, patients will receive monthly treatment up to a maximum of 6 months total.
  Other Names: Lucentis

SUMMARY:
Age Related Macular Degeneration (AMD) is the leading cause of blindness in North America. This condition causes a progressive loss of central vision, the part of your vision that allows you to read, drive and see images in sharp detail directly in front of you. The wet form of AMD is characterized by the growth and leakage of small blood vessels into the choroid layer of the eye, or the back of the eye. These leaking blood vessels disrupt the structure and function of the eye, causing loss of vision, particularly the sharp vision created by the macula area of the eye.

Currently, the best treatment for wet AMD is a series of injections of an anti-vascular endothelial growth factor (anti-VEGF) drug, ranibizumab (Lucentis). The clinical response to treatment is varied. Approximately 70% of patients see a moderate vision gain (3-line gain on a visual acuity chart), but there are 30% who do not see a similar improvement in vision. There is no way to identify those patients who will respond with significant vision gain versus those who will not experience moderate vision gain. Recent research into AMD has demonstrated that genetic mutations are proving to be key risk factors for patients developing wet AMD, with up to 80% of wet AMD cases explained by inherited genetic variations. Scientists have theorized that there may be a genetic difference between those patients who see significant responses to treatment and those who do not. The investigators will be testing participant's genetic profile using the Macula Risk test and following their progress through the standard treatment for wet AMD over the course of this study. This study aims to demonstrate the association between known genetic variations and patient responses to treatment.

DETAILED DESCRIPTION:
Your ophthalmologist will determine your suitability for this study through a screening protocol. You will have measurements of your visual acuity and will undergo a series of imaging tests as described in the next paragraph to show presence of blood vessel growth in the back of your eye (the choroid). You cannot be included in this study if you have another significant eye disease that affects your vision, if you have blood vessel growth in the back of your eye (choroid) for reasons other than AMD, if you have medically uncontrolled glaucoma, if you have been treated for AMD in that past, if you have had intra-ocular surgery in the study eye in the past 3 months, if you have had any past retinal or vitreous surgery, or if you have physical or mental disabilities that would prevent accurate vision testing.

At the beginning of the study, we will take a sample of cells from the inside of your cheek, using a small swab. The sample will be sent to a genetic laboratory for analysis and storage. This information will be kept masked for the duration of the study, meaning that you, the study ophthalmologist and the data analyzer will not know the results of the genetic test until the study is completed.

You will be asked to come in for an initial assessment to determine your starting visual abilities and medical history. On your next appointment, you will receive your first treatment of intra-vitreal injections of Ranibizumab (Lucentis). You will be asked to come into the clinic every month for six (6) months total for treatment injections and testing. At each appointment, we will take 3-D images of your retina (the back of your eye) using an Optical Coherence Tomography (OCT) imaging device, test your eye pressure and determine if there are any signs of infection or inflammation from the injections. On months 1, 3, and 6 we will also test your vision, your contrast sensitivity using a standard contrast sensitivity chart (The Pelli-Robson chart) and take images of the blood vessel growth using a coloured dye (fluorescein) to help us see your vessels. Before every treatment, anesthetic eye drops (proparacaine) will be applied to your eye so you will not feel the injections. You will be given antibiotic eye drops (Zymar®) that you will be asked to use 4 times a day for a few days after the injection to prevent infection.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be at least 18 years of age
* Choroidal neovascularization (CNV) secondary to age-related macular degeneration
* CNV under geometric center of the foveal avascular zone
* Evidence of activity on fundus fluorescein angiography
* Evidence of CNV activity as suggested by one of the following: sub-retinal hemorrhage, sub-retinal lipid, documented loss of 3 lines of vision within the last 3 months
* Visual acuity of between 20/40 and 20/300 in the study eye tested via Early treatment of Diabetic Retinopathy Study (ETDRS) eye chart score of 34 to 73 letters at 2 meters.

Exclusion Criteria:

* Individuals with choroidal neovascularization from causes other than AMD
* Patients physically unable to tolerate intravenous fluorescein angiography
* Patients with medically uncontrolled glaucoma
* Any intraocular surgery within 3 months in the study eye
* Prior retinal or vitreous surgery including vitrectomy or scleral buckling
* Any significant ocular disease other than AMD that has compromised or could compromise vision in the study eye and confound analysis of the primary outcome
* Individuals with physical or mental disabilities that prevent accurate vision testing
* History of any laser treatment of CNV in study eye (laser photocoagulation or prior photodynamic therapy), or anti-VEGF (ranibizumab or bevacizumab) in the past 6 months in the study eye.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2012-01; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Gains in visual acuity | Baseline and months 1, 2, 3, 4, 5, and 6
  Percent probability gains in visual acuity will be assessed by comparing best corrected visual acuity at each follow up appointment by the standardized vision testing, early treatment diabetic retinopathy study (ETDRS) test. The ETDRS visual acuity test was first developed to effectively evaluate visual changes following panretinal photocoagulation in patients with diabetic retinopathy. This method of measuring visual acuity was more accurate than previous methods, and thus has become the global standard, especially for clinical trials where it is essential to have utmost accuracy.

SECONDARY OUTCOMES:
Changes in choroid vessel activity in lesion growth and activity at choroid | Baseline and months 1, 2, 3, 4, 5 and 6
  The changes in blood vessel lesion growth and activity will be measured by OCT (Ocular Coherence Tomography) and fundus fluoroscein angiography to assess choroidal neovascular leakage
Rate of cataract progression | Baseline and months 1, 2, 3, 4, 5, and 6
  Measured at each appointment with a slit lamp examination
Resolution of macular edema | Baseline and months 1, 2, 3, 4, 5, 6
  The speed at which macular edema resolves will be visually measured using optical coherence tomography
Mean change in visual acuity according to identified genetic mutations | Baseline and Months 1, 2, 3, 4, 5, 6
  Mean change in visual acuity according to individual mutations at the CFH haplotypes/C3 rs2230199 marker/ARMS2 rs10490924 marker and mt A4917G marker, calculated using the Macula Risk findings and visual acuity results as determined using ETDRS visual screening
Mean change in visual acuity regardless of genetic profile results | Baseline and Months 1, 2, 3, 4, 5, 6
Interaction of smoking status and genetic profile on visual acuity changes | Baseline and Months 1, 2, 3, 4, 5, 6

CONTACTS AND LOCATIONS:
Overall Officials: Varun Chaudhary, MD, FRCSC, Principal Investigator — St. Joseph's Healthcare Hamilton/McMaster University
Locations (2):
- Canada (2):
  - St. Joseph's Healthcare Hamilton Regional Eye Centre, Hamilton, Ontario
  - Toronto Western Hospital Eye Clinic, Toronto, Ontario